CLINICAL TRIAL: NCT05751018
Title: Phase II Clinical Study of Pyrotinib in First-line Treatment of Primary HER2-amplified/Mutated Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-3350D
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pyrotinib (Experimental)
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib maleate is a small molecule tyrosine kinase inhibitor that can irreversibly inhibit HER1, HER2, and HER4.

SUMMARY:
This is a multicenter, single-arm phase II clinical study to evaluate the safety and efficacy of pyrotinib maleate as a first-line treatment for HER2-mutated or amplified non-small cell lung cancer. Pyrotinib maleate is a small molecule tyrosine kinase inhibitor that can irreversibly inhibit HER1, HER2, and HER4.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: ≥18 years old; 2. Histologically confirmed stage IIIB or IV non-small cell lung cancer; 3. Have not previously received systemic anticancer therapy for stage IIIB or IV NSCLC; 4. HER2 insertion mutation, primary HER2 point mutation or primary HER2 amplification confirmed by genetic testing of tumor tissue or blood, pleural effusion, cerebrospinal fluid and other specimens; 5. There is at least one measurable lesion determined based on RECIST 1.1; 6. ECOG score 0-1 points; 7. Expected survival period ≥ 12 weeks; 8. Cardiac ultrasound examination showed that left ventricular ejection fraction (LVEF) ≥ 50%; 9. The patient's bone marrow function, liver and kidney function were confirmed to meet the following requirements by laboratory tests before the first administration:

  1. Neutrophil count (ANC) ≥ 1,500/mm3 (1.5×109/L);
  2. Platelet count (PLT) ≥ 75,000/mm3 (75×109/L);
  3. Hemoglobin (Hb) ≥ 8 g/dL (80 g/L);
  4. Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 60 mL/min;
  5. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);
  6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤ 2.5 times the upper limit of normal (ULN), patients with liver metastases should be ≤ 5×ULN.

     10. The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

     Exclusion Criteria:
* 1. Previous use of EGFR TKI therapy; 2. Participated in clinical trials of other drugs within 4 weeks before the start of the study; 3. Symptomatic brain metastases or meningeal metastases; 4. Insufficient bone marrow reserve or insufficient organ function; 5. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow drugs, etc., may affect the intake, transport or absorption of drugs; 6. Received major surgical operation or severe traumatic injury, fracture, or poor healing wound within 4 weeks; 7. Known history of other malignancies, unless the subject has received potentially curative therapy prior to initiation of therapy and has at least 3 years of evidence of disease-free recurrence (non-small cell lung cancer, radical skin basal cell undergoing successful resection) carcinoma, superficial bladder cancer, squamous cell carcinoma of the skin, cervical carcinoma in situ or other carcinoma in situ); 8. Those who have serious adverse reactions and allergies to the drugs and excipients used in this group; 9. Pregnant or lactating female patients, female patients with fertility and positive baseline pregnancy test, or patients of childbearing age who are unwilling to take effective contraceptive measures throughout the trial; 10. The patient has serious concomitant diseases, or any other condition that the investigator considers the patient unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 year
  It is defined as the proportion of patients whose tumors shrink to a predetermined size and maintain a minimum time limit. It includes the cases of CR and PR.

SECONDARY OUTCOMES:
PFS | 1 year
  From the date Into this study to tumor progression or death for any
DCR | 2 year
  the rate of CR, PR plus SD
AEs and SAEs | 1 year
  Number of Participants With adverse events (AEs) and serious adverse events (SAEs) Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.
QoL | 1 year
  The quality of life of the subjects was assessed according to the EORTC QLQ-C30 quality of life questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College, Beijing, Beijing Municipality, China